CLINICAL TRIAL: NCT07044986
Title: Ultrasonographic Evaluation of the Ulnar Nerve in Individuals With and Without Generalized Joint Hypermobility
Status: Not yet recruiting | Type: Observational
Sponsor: Beylikduzu State Hospital (Other)
Responsible Party: Principal Investigator, Busra Sirin, Principle Investigator, Beylikduzu State Hospital
Other Study IDs: BeylikduzuStateH21
Record Dates: First submitted 2025-06-22; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Hypermobility, Joint
MeSH Terms: conditions — Joint Instability

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hypermobility: patients with generalized joint hypermobility snyndrome
  Interventions: Other: no intervention
- Control group: healthy control
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This study will include 30 individuals diagnosed with Generalized Joint Hypermobility (GJH) based on the Beighton score and 30 healthy controls without GJH. Participants will undergo Tinel's test and the flexion-compression test. The presence of ulnar nerve-related symptoms such as pain and numbness will be recorded. Ultrasonographic evaluation of the ulnar nerve will be performed at the level of the medial epicondyle, as well as 2 cm proximal and distal to it. Cross-sectional area and diameter of the ulnar nerve will be measured at each site, repeated three times, and the average will be used. Additionally, ulnar nerve mobility during elbow flexion and extension will be assessed. The nerve will be classified as stable if it remains within the cubital tunnel, subluxated if it moves to the level of the epicondyle, and dislocated if it shifts anterior to the medial epicondyle.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 40 years
* A Beighton score of 4 or higher (indicative of Generalized Joint Hypermobility)
* Willingness to participate in the study

Exclusion Criteria:

* Being under 18 or over 40 years of age
* History of surgery or fracture in the elbow region
* Presence of active infection at the measurement site
* Presence of congenital anomaly in the upper extremity
* History of surgery involving neural structures in the upper extremity
* Presence of malignancy
* Pregnancy
* Presence of cognitive or psychiatric disorders

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: hypermobility and healthy controls
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Ulnar nerve cross-sectional area (CSA) at the medial epicondyle | 0 day
  CSA measurement provides insight into nerve thickening, which may indicate entrapment or irritation.
Ulnar nerve cross-sectional area (CSA) at the 2 cm proximal of medial epicondyle | 0 day
  CSA measurement provides insight into nerve thickening, which may indicate entrapment or irritation.
Ulnar nerve cross-sectional area (CSA) at the 2 cm distal of medial epicondyle | 0 day
  CSA measurement provides insight into nerve thickening, which may indicate entrapment or irritation.
Ulnar nerve diameter | 0 day
  Ulnar nerve diameter with ultrasonography
Ulnar nerve mobility classification during elbow flexion (stable/subluxated/dislocated) | 0 day
  Dynamic USG evaluation allows visualization of nerve movement and instability during joint motion.

SECONDARY OUTCOMES:
Presence of ulnar nerve-related symptoms: | 0 day
  Symptom inquiry helps correlate clinical complaints with sonographic findings.

CONTACTS AND LOCATIONS:
Locations (1):
- Beylikdüzü State Hospital, Istanbul, Beylikdüzü, Turkey (Türkiye)